CLINICAL TRIAL: NCT03040089
Title: Efficacy and Safety of Picosecond, Neodymium-doped Yttrium Aluminum Garnet Laser Laser Therapy Using 1,064 nm and 595 nm on Patients With Melasma: A Prospective, Multi-center, Split Face, 2% Hydroquinone Cream-controlled Clinical Trial
Brief Title: Efficacy and Safety of Picosecond, Neodymium-doped Yttrium Aluminum Garnet Laser Therapy Using 1,064 nm and 595 nm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CynosureLutronic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LTN-03
Record Dates: First submitted 2017-01-24; First posted 2017-02-02 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2017-01

CONDITIONS: Melasma
MeSH Terms: conditions — Melanosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- picosecond laser & 2% hydroquinone cream (Experimental): PICO+4 laser system and Neoquine Cream 2% (2% hydroquinone cream) for melasma
  Interventions: Device: PICO+4; Drug: Neoquine Cream 2%
- 2% hydroquinone cream (Sham Comparator): Only Neoquine Cream 2% (2% hydroquinone cream) for melasma
  Interventions: Drug: Neoquine Cream 2%

INTERVENTIONS:
Device: PICO+4 — picosecond, neodymium-doped yttrium aluminum garnet laser
  Arms: picosecond laser & 2% hydroquinone cream
Drug: Neoquine Cream 2% — 2% hydroquinone cream

SUMMARY:
This is a prospective, multi-center, split-face, controlled clinical trial that aims to investigate the efficacy and safety of picosecond, neodymium-doped yttrium aluminum garnet laser laser therapy on patients with melasma, compared with 2% hydroquinone cream. The trial will be performed by two Korean institutions on 45 subjects.

ELIGIBILITY:
Inclusion Criteria:

* Females between the ages of 19 and 74
* Has Fitzpatrick Skin Type III-V
* Diagnosed with moderate to severe (GSS ≧ 2) melasma lesions
* Agreed to the prohibition of the use of local/systemic corticosteroids or retinoids and other local/systemic lightening medications, and willing to abide by such instructions
* Agreed to use the same facial skin care products during the clinical trial period (including the follow-up period), and willing to abide by such instructions
* Agreed to the daily use of an over SPF 50 sunblock on their face during the clinical trial period (including the follow-up period), and willing to abide by such instructions
* Agreed to have their face photographed
* (In case of fertile women) Tested negative in the pregnancy test and agreed to use birth control contraceptives during the clinical trial period

  * Oral contraceptives are forbidden as they may influence the results of the clinical study.
* Agreed not to undergo any other procedure on their face during their participation in the clinical trial
* Voluntarily agreed to sign the written consent form and willing to follow the instructions of the study protocol

Exclusion Criteria:

* Participated in another medical device or medication clinical trial in the last 3 months, or planning to participate in another trial during this trial
* Received a cosmetic treatment such as laser, light therapy, or surgery in their facial area in the last 6 months, or have a history of filler treatments using collagen, hyaluronic acid, or any other material
* Diagnosed with incurable melisma
* Has a history of allergic reaction to local anesthesia
* Has a history of malignant tumors on their face
* Has skin lesions such as cuts, wounds, or injuries on their face
* Pregnant or breastfeeding
* Has an infection, dermatitis, or rash on their face
* Currently diagnosed with uncontrolled diabetes or a cardiac disorder such as resistant hypertension
* Currently diagnosed with anticoagulant disease or taking anticoagulants
* Has a history of keloid scarring, hypertrophic scarring, or abnormal would healing
* Has a history of immunodeficiency or intake of immunosuppressants
* Has a history of leukoplakia, eczema, or psoriasis
* Has a history of connective tissue diseases such as systemic lupus erythematosus or scleroderma
* Has a history of convulsive disorder caused by light
* Has a history of diseases irritated by heat on their face (e.g., herpes simplex or herpes zoster)
* Has a history of radiotherapy or anticancer chemotherapy on their face
* Has a history of hormonal therapy in the last 3 months (e.g., estrogen, progesterone, or oral contraceptive)
* Has a history of use of a lightening medication (hydroquinone, tranexamic acid), isotretinoid (or retinoid), light-sensitive medication, or steroids in the last 6 months
* Has excessive facial tanning
* Other subject assessed as inadequate for the clinical trial by the investigators

Ages: 19 Years to 74 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-03-09 (Actual); Primary Completion 2016-07-15 (Actual); Study Completion 2016-09-26 (Actual)

PRIMARY OUTCOMES:
Success rate of treatment according to RL*I | Baseline, 1 week after final treatment
  The success rate is determined by the change rate (%) of the relative lightness measured before the treatment (day of screening) and 1 week after the final treatment.

SECONDARY OUTCOMES:
Relative skin lightness using the colorimeter(RL*I) | Baseline, 1 week, 4 weeks, and 12 weeks after the final treatment
mMASI (modified Melasma Area Severity Index) evaluation | Baseline, 1 week, 4 weeks, 8 weeks, and 12 weeks after the final treatment
Subject satisfaction (5-point scale questionnaires on subject's satisfaction) | 1 week and 12 weeks after the final treatment

CONTACTS AND LOCATIONS:
Overall Officials: Wonserk Kim, Principal Investigator — Kangbuk Samsung Hospital

IPD SHARING:
Plan to Share IPD: No